CLINICAL TRIAL: NCT04321044
Title: Genetic Based Analysis of Identifying Predictors of Blood Pressure Response in Hypertensive Patients After Renal Denervation
Brief Title: Genetic Based Analysis in Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Roland E. Schmieder, Full Professor of Medicine, University of Erlangen-Nürnberg Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CRC2019GBA
Record Dates: First submitted 2020-02-17; First posted 2020-03-25 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Hypertension; Renal Denervation; Genetic Predisposition
Keywords: Renal denervation; Arterial hypertension
MeSH Terms: conditions — Hypertension; Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Renal Denervation (Other): We attempt to identify predictors of blood pressure response to renal denervation by using a GWAS (Genome wide association study) approch
  Interventions: Genetic: Genetic based analysis of identifying predictors of blood pressure in patients after renal denervation

INTERVENTIONS:
Genetic: Genetic based analysis of identifying predictors of blood pressure in patients after renal denervation — We attempt to idendtify predictors of blood pressure response to renal denervation by using a GWAS (Genome wide association study) approch.

SUMMARY:
Many attempts to identify predictors of blood pressure response after renal denervation failed to identify a meaningful determination of blood pressure response.

These attempts have been based on demographic parameters, clinical parameters, endocrine inflammatory and other biochemical variables, comorbidities and disease factors. So far the only predictor of blood pressure response is the pre-treatment blood pressure. According to Wilder's law the pre-treatment baseline value is always a determinant for any change due to an intervention, irrespective which biological variable is examined.

The investigators propose a genetic approach to identify predictors of blood pressure response after renal denervation. Genetic factors are not subject to changes of clinical parameters, previous or current antihypertensive therapy, hypertension associated organ damages, comorbidities and other potential clinical variables.

DETAILED DESCRIPTION:
Background:

Up to now numerous attempts to identify predictors of blood pressure response after renal denervation failed to identify a meaningful and consistent determinant of blood pressure response. These approaches have been based on demographic parameters, clinical parameters, comorbidities and disease factors as well as numerous endocrine inflammatory and other biochemical variables. Only the pre-treatment blood pressure emerged as a predictor of blood pressure response which is no surprise since according to Wilder's law the pre-treatment baseline value is always a determinant for any change due to an intervention, irrespective which biological variable is examined, e.g. blood pressure, LDL cholesterol, HbA1c and so on.

The investigators suggest a genetic approach to identify predictors of blood pressure response after renal denervation. The rationale is quite simple: Genetic factors are not subject to changes of clinical parameters, previous or current antihypertensive therapy, hypertension associated organ damages, comorbidities, and other potential clinical variables. By such an approach the investigators previously were very successful to identify several parameters of modulators hypertensive organ damage that could not have been identified by pathophysiological or pharmaceutical maneuvers. THE INVESTIGATORS PREFER TO RUN A GENOM WIDE ASSOCIATION STUDY AND THE PARTNERS IN GLASGOW AND EDINBURGH HAVE THE DEEP KNOWLWEDGE; EXPERIENCE AND CAPACITY TO RUN A NGS (next generation sequencing, so that's the complete genome)) INCLUDING ALL BIOINFORMATICS AND OTHER ANALYSIS

Objective:

The investigators attempt to identify predictors of blood pressure response to renal denervation by using a GWAS (genome wide association study) approach. This allows to identify various suspected and unexpected polymorphism that are of interest and potentially being strong predictors of blood pressure response. By that approach the investigators will identify novel mechanism of action that are important for blood pressure response (by identifying polymorphism that are beyond the classical thinking how renal denervation may exert blood pressure lowering effects).

Study design:

In collaboration with the Homburg Group (Prof. Dr. Felix Mahfoud), the investigators will extract DNA from stored samples of patients with uncontrolled treatment resistant hypertension and perform a genome wide association study analysis (GWAS) in two cohorts: no/low responders vs. high/excellent responders. NGS will be applied by the partners in Glasgow and Edinburgh. All patients with renal denervation will be categorized according to their pretreatment adjusted blood pressure response and the investigators will compare the upper quartile vs. the lower quartile of all patients that has been so far studied in Homburg and Erlangen. By excluding those patients with a medium or average blood pressure response, the investigators will have two distinct response patterns: low/no response vs. high/excellent response.

By applying standard biostatistics analysis, the investigators will come up with a pattern of polymorphism that are significantly different between the two groups. These identified polymorphisms (or a pattern of it) may be refer, not unexpectedly, to renin angiotensin aldosterone system, sodium and water balance, sympathetic nervous system or other endocrine parameters related to hypertension. In addition to that, the investigators may find significant results of polymorphisms involved in other pathophysiologic pathways not related to hypertension (by our current knowledge) and that the Investigators have not thought about to be related to uncontrolled hypertension. These novel mechanism need to be subsequently further analyzed, but they will offer the opportunity to find novel predictors of blood pressure response.

ELIGIBILITY:
Inclusion Criteria:

* Individual is ≥ 18 and ≤ 85 years of age.
* Individual agrees to have all study procedures performed, and is competent and willing to provide written, informed consent to participate in this clinical study
* Renal denervation ≥ 6 months
* 24-h ABPM

Exclusion Criteria:

* Individual has renal artery anatomy that is ineligible for treatment including:

  1. Main renal arteries < 4 mm in diameter or < 20 mm in length.
  2. Hemodynamically or anatomically significant renal artery abnormality or stenosis in either renal artery which, in the eyes of the operator, would interfere with safe cannulation of the renal
  3. A history of prior renal artery intervention including balloon angioplasty or stenting.
  4. Multiple main renal arteries in either kidney.
* Individual has an estimated glomerular filtration rate (eGFR) of < 45mL/min/1.73m2, using the MDRD calculation.
* Individual has type 1 diabetes mellitus.
* Individual has experienced a myocardial infarction, unstable angina pectoris, or a cerebrovascular accident within 6 months of the screening visit, or has widespread atherosclerosis, with documented intravascular thrombosis or unstable plaques.
* Individual has a scheduled or planned surgery or cardiovascular intervention in the next 6 months.
* Individual has hemodynamically significant valvular heart disease for which reduction of blood pressure would be considered hazardous.
* Individual has an implantable cardioverter defibrillator (ICD) or pacemaker, or any other metallic implant which is not compatible with magnetic resonance imaging (MRI).
* Individual has any serious medical condition, which in the opinion of the investigator, may adversely affect the safety and/or effectiveness of the participant or the study (i.e., patients with clinically significant peripheral vascular disease, abdominal aortic aneurysm, bleeding disorders such as thrombocytopenia, hemophilia, or significant anemia, or arrhythmias such as atrial fibrillation).
* Individual is pregnant, nursing or planning to be pregnant. [Female participants of childbearing potential must have a negative serum or urine human chorionic gonadotropin (hCG) pregnancy test prior to treatment.]
* Individual has a known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or would be unlikely or unable to comply with study follow-up requirements.
* Individual is currently enrolled in another investigational drug or device trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Identifying predictors of systolic blood pressure by 24-h ABPM | 6 months
  To identify predictors of systolic blood pressure response after renal denervation as evaluated by 24-h ABPM by using a GWA (genome wide association) approach.

SECONDARY OUTCOMES:
Identifying predictors of diastolic blood pressure by 24-h ABPM | 6 months
  To identify predictors of diastolic blood pressure response after renal denervation as evaluated by 24-h ABPM by using a GWA (genome wide association) approach.
Identifying predictors of pulse pressure by 24-h ABPM | 6 months
  To identify predictors of pulse pressure response after renal denervation as evaluated by 24-h ABPM by using a GWA (genome wide association) approach.
Identifying predictors of systolic blood pressure by office blood pressure | 6 months
  To identify predictors of systolic blood pressure response after renal denervation as evaluated by office blood pressure by using a GWA (genome wide association) approach.
Identifying predictors of diastolic blood pressure by office blood pressure | 6 months
  To identify predictors of diastolic blood pressure response after renal denervation as evaluated by office blood pressure by using a GWA (genome wide association) approach.
Identifying predictors of pulse pressure by office blood pressure | 6 months
  To identify predictors of pulse pressure response after renal denervation as evaluated by office blood pressure by using a GWA (genome wide association) approach.

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, MD, Principal Investigator — University Hospital Erlangen
Locations (3):
- Germany (2):
  - Klinik für Innere Medizin III, Kardiologie, Angiologie Und Internistische Intensivmedizin, Saarland University Hospital, Saarland University, Homburg, Saarland
  - Clinical Research Center, Department of Nephrology and Hypertension, University of Erlangen-Nuremberg, Erlangen
- Institute of Cardiovascular and Medical Science, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Messerli FH, Bangalore S, Schmieder RE. Wilder's principle: pre-treatment value determines post-treatment response. Eur Heart J. 2015 Mar 1;36(9):576-9. doi: 10.1093/eurheartj/ehu467. Epub 2014 Dec 23. No abstract available. PMID 25540187
- [Background] Zolk O, Ott C, Fromm MF, Schmieder RE. Effect of the rs168924 single-nucleotide polymorphism in the SLC6A2 catecholamine transporter gene on blood pressure in Caucasians. J Clin Hypertens (Greenwich). 2012 May;14(5):293-8. doi: 10.1111/j.1751-7176.2012.00618.x. Epub 2012 Apr 9. PMID 22533655
- [Background] Ott C, Schneider MP, Delles C, Schlaich MP, Hilgers KF, Schmieder RE. Association of (pro)renin receptor gene polymorphism with blood pressure in Caucasian men. Pharmacogenet Genomics. 2011 Jun;21(6):347-9. doi: 10.1097/FPC.0b013e328344cdd2. PMID 21346687
- [Background] Ritt M, Ott C, Delles C, Schneider MP, Schmieder RE. Impact of the endothelial nitric oxide synthase gene G894T polymorphism on renal endothelial function in patients with type 2 diabetes. Pharmacogenet Genomics. 2008 Aug;18(8):699-707. doi: 10.1097/FPC.0b013e32830500b1. PMID 18622262
- [Background] Ott C, Schwarz T, Hilgers KF, Kreutz R, Schlaich MP, Schmieder RE. Left-ventricular structure and function are influenced by angiotensinogen gene polymorphism (-20 A/C) in young male patients. Am J Hypertens. 2007 Sep;20(9):974-80. doi: 10.1016/j.amjhyper.2007.03.008. PMID 17765139
- [Background] Ott C, Titze SI, Schwarz TK, Kreutz R, Hilgers KF, Schmidt BM, Schlaich MP, Schmieder RE. High sodium intake modulates left ventricular mass in patients with G expression of +1675 G/A angiotensin II receptor type 2 gene. J Hypertens. 2007 Aug;25(8):1627-32. doi: 10.1097/HJH.0b013e3281cd40f5. PMID 17620959
- [Background] Zolk O, Jacobi J, Pahl A, Fromm MF, Schmieder RE. MDR1 genotype-dependent regulation of the aldosterone system in humans. Pharmacogenet Genomics. 2007 Feb;17(2):137-44. doi: 10.1097/01.fpc.0000239969.46594.d0. PMID 17301693
- [Background] Fromm MF, Schmidt BM, Pahl A, Jacobi J, Schmieder RE. CYP3A5 genotype is associated with elevated blood pressure. Pharmacogenet Genomics. 2005 Oct;15(10):737-41. doi: 10.1097/01.fpc.0000175599.49764.98. PMID 16141800
- [Background] Hilgers KF, Delles C, Veelken R, Schmieder RE. Angiotensinogen gene core promoter variants and non-modulating hypertension. Hypertension. 2001 Dec 1;38(6):1250-4. doi: 10.1161/hy1201.096545. PMID 11751698
- [Background] Delles C, Erdmann J, Jacobi J, Hilgers KF, Fleck E, Regitz-Zagrosek V, Schmieder RE. Aldosterone synthase (CYP11B2) -344 C/T polymorphism is associated with left ventricular structure in human arterial hypertension. J Am Coll Cardiol. 2001 Mar 1;37(3):878-84. doi: 10.1016/s0735-1097(00)01174-8. PMID 11693765
- [Background] Schmieder RE, Erdmann J, Delles C, Jacobi J, Fleck E, Hilgers K, Regitz-Zagrosek V. Effect of the angiotensin II type 2-receptor gene (+1675 G/A) on left ventricular structure in humans. J Am Coll Cardiol. 2001 Jan;37(1):175-82. doi: 10.1016/s0735-1097(00)01063-9. PMID 11153734